CLINICAL TRIAL: NCT06117839
Title: Comparative Study Between Rate of Infection After Using Antibiotic Loaded Cement and Regular Cement in Total Knee Arthroplasty
Brief Title: Rate of Infection After Using Antibiotic Loaded Cement and Regular Cement in Total Knee Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Sallam Abo El-azaiem Mohamed, Resident physcian at orthopedic surgery and truamatology, Assiut University
Other Study IDs: ahmedsallam
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Primary Osteoarthritis of Knee Nos

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: first group is patients will be treated with regular bone cement . Patients will be routinely monitored for clinical signs of infection, including cellulitis or draining sinuses. Radiographs were obtained at 2,6 and 12 months.
  * Laboratory tests as CRP and CBC will beused to assess the infection.
  * A negative CRP indicate clean field .
  Interventions: Procedure: using antibiotic loaded cement and regular cement after total knee arthroplasty in primary knee osteoarthritis.
- 2: the second one is patient will be treated with antibiotic loaded bone cement, commonly used antibiotic includeGentamycin powder.
  Patients will beroutinely monitored for clinical signs of infection, including cellulitis or draining sinuses. Radiographs were obtained at 2,6 and 12 months.
  * Laboratory tests as CRP and CBC used to assess the infection.
  * A negative CRP indicate clean field.
  Interventions: Procedure: using antibiotic loaded cement and regular cement after total knee arthroplasty in primary knee osteoarthritis.

INTERVENTIONS:
Procedure: using antibiotic loaded cement and regular cement after total knee arthroplasty in primary knee osteoarthritis. — -There are 2 groups ,first group is patients will betreated with regular bone cement ,the second one is patient will be treated with antibiotic loaded bone cement, commonly used antibiotics include Gentamycin powder .

SUMMARY:
Our study will be a prospective study To compare between the rate of infection after using antibiotic loaded cement and regular cement after total knee arthroplasty in primary knee osteoarthritis.this will be at assiut university trauma hospital .There are 2 groups ,first group is patients will be treated with regular bone cement ,the second one is patient will be treated with antibiotic loaded bone cement, commonly used antibiotics includeGentamycin powder.

DETAILED DESCRIPTION:
Total Joint arthroplasty (TJA) is among the major and most successful orthopedic surgeries . It is indicated when there is impaired joint function that requires prosthesis replacement .Total hip arthroplasty (THA) and total knee arthroplasty (TKA) are the most replaced joints . TKA is becoming more common over the world, with 5 million degenerative knee joint replacement procedures projected by 2030 .

Although perioperative antimicrobial procedures have improved significantly, periprosthetic joint infection (PJI) following TKA remains a serious complication for patients and a significant burden on the healthcare system . PJI is a leading cause of TKA revision surgery, accounting for more than 15% of all revisions.that can cause a long hospital stay, increase the risk of readmission, and lead to poor patient outcomes, such as decreased function and a lower quality of life. In the worst case, PJI can lead to amputation or even death .

Antibiotic-loaded bone cement (ALBC) has been recommended to reduce the risk of PJI. The aim of such a strategy is to promptly release antibiotics at the action site with very little systemic exposure, which may not be achieved by systemic antibiotics due to insufficient blood supply (1) but in the literature, it is uncertain whether ALBC or plain bone cement (PBC) should be used in PTKA. ALBC has been shown to decrease significant complications, although it has the disadvantage of diminishing cement strength. A meta-analysis published in 2015 discovered no statistically significant difference in the incidence of PJI in patients receiving two cement materials during PTKA , another meta-analysis was done in 2022 demonstrated that the preventive application of ALBC during PTKA could reduce the rates of deep PJI, However, the existing related articles are mostly single-center and retrospective studies, and further high-quality ones are needed for confirmation ,so we will conduct our study to compare between ALBC and PBC in TKA infection.

ELIGIBILITY:
Inclusion Criteria:

* Patient with primary knee osteoarthritis.
* Patient underwent total knee arthroplasty.

Exclusion Criteria:

* Patient with rheumatoid knee osteoarthritis.
* Patient with post-traumatic knee osteoarthritis.
* Patient with knee tumor.
* Patient has allergy to antibiotics used in the study.
* Patient with any operative procedure in the knee.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patient undergo TKA in primary osteoarthritis. Patient with rheumatoid knee osteoarthritis.
  Patient with post-traumatic knee osteoarthritis, Patient with knee tumor. Patient has allergy to antibiotics used in the study or Patient with any operative procedure in the knee are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Infection eradication rate | 12 months postoperative
  patients will be evaluated clinically and undergo lab evaluation (CRP and CBC).Patients will be routinely monitored for clinical signs of infection, including cellulitis or draining sinuses. Radiographs will be obtained at 2,6 and 12 months.
  * Laboratory tests as CRPwill be used to assess the infection.
  * A negative CRP indicate clean field and eradication of infection.

SECONDARY OUTCOMES:
Cost/benefit ratio. | 12 months postoperative
  study the cost in egyptian pound